CLINICAL TRIAL: NCT03192202
Title: Clinical and Biological Evaluation of the Novel CD30/CD16A Tetravalent Bispecific Antibody (AFM13) in Relapsed or Refractory CD30-Positive Lymphoma With Cutaneous Presentation: A Biomarker Phase Ib/IIa Study
Brief Title: AFM13 in Relapsed/Refractory Cutaneous Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ahmed Sawas (Other)
Responsible Party: Sponsor-Investigator, Ahmed Sawas, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAP4461
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Lymphoma, T-Cell, Cutaneous
Keywords: Lymphoma; Cutaneous Lymphoma; cutaneous T-cell lymphoma (CTCL); CD30-Positive Cutaneous Lymphoma; T-cell lymphoma; PTCL; CTCL; CD30; immunotherapy
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma; Lymphoma, T-Cell | interventions — AFM13

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 1.5 mg/kg of AFM13 once weekly for weeks 1-8.
  Interventions: Drug: AFM13
- Cohort 2 (Experimental): 7 mg/kg of AFM13 once weekly for weeks 1-8.
  Interventions: Drug: AFM13
- Cohort 3 (Experimental): 7mg/kg CIVI for weeks 1-8.
  Interventions: Drug: AFM13
- Cohort 4 (Experimental): 200mg flat dose once weekly for 8 weeks.
  Interventions: Drug: AFM13

INTERVENTIONS:
Drug: AFM13 — AFM13 is a recombinant antibody construct against human CD30 and CD16A. It will be given to patients intravenously at the dose and schedule applicable to the cohort the patient was enrolled in specified in the various arms listed.
  Other Names: AFM13 recombinant antibody

SUMMARY:
The investigators plan to investigate AFM13 and evaluate its ability to facilitate and redirect the Natural Killer (NK) cells in eliminating CD30-positive lymphoma targets in the skin and, by inference, other organs involved by the lymphoma.

DETAILED DESCRIPTION:
This is an open label, Phase Ib/IIa study designed to evaluate the biologic activity of AFM13 in patients with relapsed or refractory CD30-positive lymphomas with cutaneous involvement. Primary cutaneous CD30-positive lymphoproliferative disorders (LPD) represent a spectrum from lymphomatoid papulosis (LyP), to primary cutaneous anaplastic large cell lymphoma (C-ALCL), to transformed mycosis fungoides (TMF).

The most indolent form of primary cutaneous CD30-positive LPD is LyP, which is usually well controlled with low dose oral methotrexate, but control of the disease frequently requires life-long therapy. In contrast, TMF is an aggressive disease which does not have a standard of care, as patients are treated with various modalities of care with variable outcomes). The spectrum of other CD30-positive lymphomas with cutaneous presentation is very broad and involves systemic B and T cell lymphomas with various clinical behaviors.

Redirecting Natural Killer (NK) cells towards these CD30-positive malignancies through direct engagement with AFM13 is expected to induce tumor cell killing through NK cell-mediated and T cell-mediated cytotoxicity (i.e., cytotoxic T lymphocytes (CTL)).

The primary objective of this trial is to study the biologic and immunologic effects induced by the administration of various doses of AFM13, when given as a single agent.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed CD30-positive lymphoma with cutaneous involvement
* Failure or intolerance to at least one prior therapy for the current disease
* Presence of one or more cutaneous lesions (measuring at least 1 cm x 1 cm in size; if only one lesion is present it should be up to the investigator discretion to determine eligibility)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate organ and marrow function
* Platelets ≥50,000/μL
* Absolute neutrophil count ≥ 1,000/μL
* Bilirubin < 1.5 x institutional upper limit of normal (ULN) or < 3 x ULN in patients with Gilbert's disease or liver involvement
* Serum albumin ≥ 2.0 g/dL
* Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤2.5 × institutional ULN or, in the case of liver involvement by the primary disease AST/ALT ≤ 5 x ULN
* Creatinine≤1.5 x institutional ULN or estimated creatinine clearance of ≥45 mL/min by the Cockcroft-Gault equation or measured creatinine clearance >45 mL/min
* Females of child bearing potential must have a negative serum pregnancy test with 7 days prior to first dose of treatment. Female patients of childbearing potential and all male partners must agree to use double barrier methods of contraception throughout the study period and for at least 30 days following investigational product discontinuation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Any cancer-related therapy for the current disease within 2 weeks of screening (all supportive care measures are allowed)
* Major surgery within 2 weeks prior to first dose of study drug
* Evidence of active central nervous system (CNS) involvement
* Requirement for systemic immunosuppressive therapy (e.g. Graft-versus-Host Disease (GVHD) therapy within 12 weeks before the first dose of study drug)
* Uncontrolled concurrent serious illness.
* Concurrent malignancy or history of a previous malignancy within 3 years prior to first dose of the current study, unless curatively resected basal, squamous cell carcinoma of the skin, or cervical carcinoma in situ.
* Active infections including hepatitis B carrier status, hepatitis C virus (HCV) infection (patients must have a negative Hepatitis B and Hepatitis C viral load at screening)
* Known HIV-positive status
* Any significant medical conditions, laboratory abnormality, or psychiatric illness that would exclude the subject from participation or interfere with study treatment, monitoring and compliance such as:
* unstable angina pectoris, symptomatic congestive heart failure (New York Heart Association (NYHA) III or IV), myocardial infarction ≤ 6 months prior to first study drug, clinically significant and uncontrolled cardiac arrhythmia (e.g. atrial fibrillation/flutter ventricular cardiovascular physiology is allowed), cerebrovascular accidents ≤ 6 months before study drug start
* severely impaired lung function
* Serious, systemic infection requiring treatment ≤7 days before the first dose of study drug
* Any severe, uncontrolled disease or condition which in the investigator's opinion, may put the subject at significant risk, may confound the study results, or impact the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Sawas, MD, Principal Investigator — Columbia University
Locations (1):
- Center for Lymphoid Malignancies, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2: 7.0 mg/kg of AFM13 once weekly for weeks 1-8.
  AFM13: AFM13 is a recombinant antibody construct against human CD30 and CD16A. It will be given to patients intravenously at the dose and schedule applicable to the cohort the patient was enrolled in specified in the various arms listed.
- Cohort 3: 7.0 mg/kg CIVI of AFM13 once weekly for weeks 1-8.
  AFM13: AFM13 is a recombinant antibody construct against human CD30 and CD16A. It will be given to patients intravenously at the dose and schedule applicable to the cohort the patient was enrolled in specified in the various arms listed.
- Cohort 4: 200 mg ( Flat dose) of AFM13 once weekly for weeks 1-8.
  AFM13: AFM13 is a recombinant antibody construct against human CD30 and CD16A. It will be given to patients intravenously at the dose and schedule applicable to the cohort the patient was enrolled in specified in the various arms listed.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 3 | 3 | 3 | 6
Completed | 3 | 3 | 3 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 5 | 12
  >=65 years | 1 | 0 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 5
  Male | 2 | 2 | 2 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 2 | 6
  White | 3 | 1 | 1 | 4 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Incidence of Treatment-Emergent Adverse Events [Safety and Toxicity] broken down by adverse event and CTCAE v4.0 grade of each event.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants
  G3/4 Infection and skin rash | 1 | 0 | 0 | 0
  G1 IRR | 0 | 2 | 0 | 0
  Death, G3 infection , IRR | 0 | 1 | 0 | 0
  No AE | 2 | 0 | 3 | 6

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The sum of patients with partial responses and complete responses.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1; Cohort 3: 2/3 responses
- Cohort 2: No response
- Cohort 4: 2/6 responders
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 2 | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 3/3 | 0/3 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=6)
G3/4 Infection and skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 | 0
G1 IRR (General disorders) | 0 (0) | 1 (1) | 0 | 0
Death, G3 infection, IRR (General disorders) | 0 | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=6)
Infusion related reaction (IRR) (General disorders) | 0 (0) | 3 (12) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03192202/Prot_SAP_000.pdf